CLINICAL TRIAL: NCT04719182
Title: Practice of Adjunctive Treatments in Intensive Care Unit Patients With Coronavirus Disease 2019 (PRoAcT-COVID) - an Observational Study in the Netherlands
Brief Title: Practice of Adjunctive Treatments in Intensive Care Unit Patients With COVID-19
Acronym: PRoAcT-COVID
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof. Dr. Marcus J. Schultz, Prof., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: PRoAcT-COVID
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Covid19; Pneumonia; Thrombosis; Thromboembolism; Anticoagulants; Increased; ARDS, Human
Keywords: ARDS; COVID-19; Lungembolism; DVT; PPI; Adjunctive therapies; Mechanical ventilation; Prone positioning
MeSH Terms: conditions — COVID-19; Pneumonia; Thrombosis; Thromboembolism; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Adjunctive therapies — Determine and compare practice of adjunctive and supportive treatments for COVID-19

SUMMARY:
Rationale Many patients with coronavirus disease (COVID-19) need hospital admission for oxygen supplementation. A substantial number of patients need intensive care unit (ICU) admission for escalation of care. ICU doctors and nurses are struggling to provide the best care for patients with COVID-19. Practice of adjunctive and supportive treatments remains uncertain.

Objective To determine and compare practice of adjunctive and supportive treatments for COVID-19 in the Netherlands, and to determine their independent associations with outcome.

Hypotheses Practice of adjunctive and supportive treatments for COVID-19 varies substantially. Adjunctive and supportive treatments have an independent association with outcome in ICU patients with COVID-19.

Study design National/international, multicenter, retrospective observational study. Study population Intensive care unit (ICU) patients with COVID-19.

Methods In this study we will collect data on diverse treatments during the first 28 days in ICU, including (a) the types of oxygen support* and awake prone positioning; (b) the types of ventilatory support, (c) rescue therapies for refractory hypoxemia during invasive ventilation (prone positioning, ventilator adjustments, continuous muscle paralysis, and extracorporeal membrane oxygenation); (d) adjunctive treatments, including thromboprophylaxis and anticoagulation, antiviral and immunomodulating therapies, and (e) experimental supportive treatments. Outcomes include duration of each adjunctive treatment, duration of ventilation, incidence of tracheostomy, duration of stay in ICU and mortality until day 90.

Study endpoints A combination of adjunctive treatments, including types of oxygen support, ventilatory support and rescue therapies for refractory hypoxemia during invasive ventilation (primary), other adjunctive and supportive treatments, tracheostomy rate; duration of ventilation and ventilator-free days and alive at day 28 (VFD-28), duration of ICU and hospital stay, and ICU, hospital and 90-day mortality.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness Retrospective collection of data regarding adjunctive treatments, and clinical endpoints is without risk for ICU patients.

*In a subset of patients we will collect granular data (every two hours) regarding oxygenation (FiO2, inspiratory tidal volume, air flow, respiratory rate, SpO2, PaO2, and PEEP) over the first 2 full calendar days of ICU admission. The primary endpoint of this sub-analysis will be the amount of oxygen used with different respiratory support interventions. The statistical analysis plan for the analysis of these data that were collected in two ICUs that participated in the national study, and one additional ICU in Spain is uploaded in the document section (filename Statistical Analysis Plan PROXY-COVID)

ELIGIBILITY:
Inclusion Criteria:

* COVID-19, confirmed with PCR; and
* Admission to one of the participating ICUs, or an emergency location that serves as an ICU during the pandemic.

Exclusion Criteria:

* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe coronavirus disease 2019 (COVID-19) admitted to intensive care units (ICUs) in the Netherlands between September 2020 and January 2021 (i.e. during the second surge of COVID-19 patients).
Sampling Method: Non-Probability Sample
Enrollment: 1011 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Mortality | 90 days
ICU, hospital and 90-day mortality | 90 days
Ventilator-free days and alive at day 28 | 28 days
ICU length of stay | 90 days
Hospital length of stay | 90 days

SECONDARY OUTCOMES:
Proven deep vein thrombosis (DVT) | 28 days
Incidence of gastrointestinal bleeding | 28 days
Development of acute kidney injury (AKI) | 28 days
Incidence of tracheostomy | 28 days
Use of renal replacement therapy (RRT) | 28 days
Proven pulmonary embolism (PE) | 28 days

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Amsterdam UMC location AMC, Amsterdam
  - Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA), Amsterdam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van der Ven FLIM, Valk CMA, Blok S, Brouwer MG, Go DM, Lokhorst A, Swart P, van Meenen DMP, Paulus F, Schultz MJ; PRoAcT-COVID study investigators. Broadening the Berlin definition of ARDS to patients receiving high-flow nasal oxygen: an observational study in patients with acute hypoxemic respiratory failure due to COVID-19. Ann Intensive Care. 2023 Jul 14;13(1):64. doi: 10.1186/s13613-023-01161-6. PMID 37452196
- [Derived] Valk CMA, Swart P, Boers LS, Botta M, Bos LDJ, de Abreu MG, Hol L, Hollmann MW, Horn J, Martin-Loeches I, Mazzinari G, Myatra SN, Nijbroek SG, Rosenberg NM, Stilma W, Tsonas AM, van der Ven WH, Neto AS, Schultz MJ, Paulus F. Practice of adjunctive treatments in critically ill COVID-19 patients-rational for the multicenter observational PRoAcT-COVID study in The Netherlands. Ann Transl Med. 2021 May;9(9):813. doi: 10.21037/atm-21-764. PMID 34268426

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-05-18): https://cdn.clinicaltrials.gov/large-docs/82/NCT04719182/SAP_000.pdf